CLINICAL TRIAL: NCT00799981
Title: A Multi Centre, Single-blind, Randomized, Cross-over Study Comparing Two Female Catheters With Different Length in Terms of Residual Urine After Intermittent Catheterization
Brief Title: A Comparison of Two Urinary Catheters of Different Lengths for Female Use, in Intermittent Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: YA-LOF-0015
Record Dates: First submitted 2008-11-28; First posted 2008-12-01 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Catheterization

STUDY DESIGN:
Intervention Model Description: The study was designed as a randomised, single blind, cross-over study to eliminate bias.
  Every subject was catheterisized with both 7 cm and 10 cm long catheters.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The subjects were handed out numbered boxes with the catheter randomised to be used and then cathererisized by herself.
  The investigator was blinded to which catheter was used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- AABB (Experimental): A=Coloplast SpeediCath Compact catheter, 7 cm B=Astra Tech POBE catheter, 10 cm 7 cm then 7 cm then 10 cm then 10 cm
  Four catheterizations in total, two catheterizations with each study product in a randomized order.
  Interventions: Device: A=SpeediCath Compact 7 cm and B=POBE 10 cm
- ABAB (Experimental): A=Coloplast SpeediCath Compact catheter, 7 cm B=Astra Tech POBE catheter, 10 cm 7 cm then 10 cm then 7 cm then 10 cm
  Four catheterizations in total, two catheterizations with each study product in a randomized order.
  Interventions: Device: A=SpeediCath Compact 7 cm and B=POBE 10 cm
- ABBA (Experimental): A=Coloplast SpeediCath Compact catheter, 7 cm B=Astra Tech POBE catheter, 10 cm 7 cm then 10 cm then 10 cm then 7 cm
  Four catheterizations in total, two catheterizations with each study product in a randomized order.
  Interventions: Device: A=SpeediCath Compact 7 cm and B=POBE 10 cm
- BAAB (Experimental): A=Coloplast SpeediCath Compact catheter, 7 cm B=Astra Tech POBE catheter, 10 cm 10 cm then 7 cm then 7 cm then 10 cm
  Four catheterizations in total, two catheterizations with each study product in a randomized order.
  Interventions: Device: A=SpeediCath Compact 7 cm and B=POBE 10 cm
- BABA (Experimental): A=Coloplast SpeediCath Compact catheter, 7 cm B=Astra Tech POBE catheter, 10 cm 10 cm then then 7 cm then 10 cm then 7 cm
  Four catheterizations in total, two catheterizations with each study product in a randomized order.
  Interventions: Device: A=SpeediCath Compact 7 cm and B=POBE 10 cm
- BBAA (Experimental): A=Coloplast SpeediCath Compact catheter, 7 cm B=Astra Tech POBE catheter, 10 cm 10 cm then 10 cm then 7 cm then 7 cm
  Four catheterizations in total, two catheterizations with each study product in a randomized order.
  Interventions: Device: A=SpeediCath Compact 7 cm and B=POBE 10 cm

INTERVENTIONS:
Device: A=SpeediCath Compact 7 cm and B=POBE 10 cm — Catheterization should resemble the daily use as far as possible and at least 2 hours had to pass between 2 catheterizations.The study centre decided whether the subject performed all four catheterizations on one or several days.
  Other Names: Coloplast SpeediCath Compact 7 cm; Astra Tech POBE 10 cm

SUMMARY:
A study comparing a 10 cm catheter with a 7 cm catheter in a group of female patients who, on a routine bases, empty their bladder using urinary catheters, by measuring residual urine after intermittent catheterization.

DETAILED DESCRIPTION:
The study personnel will conduct three bladder scans after each catheterization in order to obtain the mean residual urine volume. Each patient will catheterize herself two times with each product, i.e. a total of four catheterizations.

Diagnosis and BMI will be collected at visit 1 to assess whether the residual urine volume differs between these subgroups.

The hypothesis that the mean residual volumes were equal when using the 7 and the 10 centimeter catheters was tested by means of the Wilcoxon signed rank test.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent
* Female subjects aged 18 years and over
* Experienced users of CIC with a minimum of one month of use
* Practice CIC a minimum of 1 time per day
* Practice CIC with female catheters with a maximum length of 20 cm
* Perform self-catheterization
* Sufficient hand function to be able to open and handle catheter packages
* Use catheters with Ch 10, 12 or 14

Exclusion Criteria:

* Pregnancy
* Ongoing symptomatic UTI
* Involvement in the planning and conduct of the study (applies to both Astra Tech staff or staff at the study site)
* Previous enrolment or randomisation of treatment in the present study
* Participation in another clinical study during the study period
* Severe non-compliance to protocol as judged by the investigator and/or Astra Tech

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Malmqvist, MD, PhD, Assoc.Prof., Principal Investigator — Clinical Research and Trial Centre, Lund University Hospital
Locations (3):
- Sweden (3):
  - Rehabiliteringskliniken, Södra Älvsborgs Sjukhus, Borås
  - Verksamhet Urologi, Sahlgrenska Universitetssjukhuset, Gothenburg
  - Clinical Research and Trial Centre, Lund University Hospital, Lund

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Each subject eligible for entry into the study was a female using catheters for intermittent self catheterization at least once a day and had done so for the last month.
  Three centers in Sweden were involved. Four catheterizations, two with each product in a randomized order, were performed at the study centre.
  Catheterization should resemble the daily use as far as possible.
Groups:
- AABB: 7 cm then 7 cm then 10 cm then 10 cm
  B=Astra Tech POBE catheter, 10 cm A=Coloplast SpeediCath Compact catheter, 7 cm
  Four catheterizations, two with each product in a randomized order.
- ABAB: 7 cm then 10 cm then 7 cm then 10 cm
  B=Astra Tech POBE catheter, 10 cm A=Coloplast SpeediCath Compact catheter, 7 cm
  Four catheterizations, two with each product in a randomized order.
- ABBA: 7 cm then 10 cm then 10 cm then 7 cm
  B=Astra Tech POBE catheter, 10 cm A=Coloplast SpeediCath Compact catheter, 7 cm
  Four catheterizations, two with each product in a randomized order.
- BAAB: 10 cm then 7 cm then 7 cm then 10 cm
  B=Astra Tech POBE catheter, 10 cm A=Coloplast SpeediCath Compact catheter, 7 cm
  Four catheterizations, two with each product in a randomized order.
- BABA: 10 cm then 7 cm then 10 cm then 7 cm
  B=Astra Tech POBE catheter, 10 cm A=Coloplast SpeediCath Compact catheter, 7 cm
  Four catheterizations, two with each product in a randomized order.
- BBAA: 10 cm then 10 cm then 7 cm then 7 cm
  B=Astra Tech POBE catheter, 10 cm A=Coloplast SpeediCath Compact catheter, 7 cm
  Four catheterizations, two with each product in a randomized order.
Period: Overall Study
Arm/Group | AABB | ABAB | ABBA | BAAB | BABA | BBAA
Started (It differs between subjects if they are catheterisized twice per visit or one catheterisation at each visit. The subjects that were catheterisized twice during one day had at least 2 hours between 2 catheterizations.) | 10 | 9 | 10 | 10 | 11 | 10
Completed | 10 | 9 | 10 | 10 | 11 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Four Catheterizations, Each Subject Was Catheterisized Twice With Each Product in a Randomized Order: A=Coloplast SpeediCath Compact catheter, 7 cm B=Astra Tech POBE catheter, 10 cm 6 arms with the following order of catheters used: AABB ABAB ABBA BAAB BABA BBAA BBAA
Arm/Group | Four Catheterizations, Each Subject Was Catheterisized Twice With Each Product in a Randomized Order
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.20 (15.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 60
Weight [Mean (Standard Deviation); unit: Kilogramme] | 66.53 (13.98)
Height [Mean (Standard Deviation); unit: Cm] | 163.62 (7.48)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.78 (4.52)

OUTCOME MEASURES:

1. Primary Outcome: Bladder Scan Measurements of Residual Urine Volume
Description: Measurements were performed with the bladder scan BVI 3000. The primary outcome variable was average residual urine volume (mL) calculated from repetitive bladder scans performed after each catheterization.
  Three bladder scan measurements were performed immediately after each catheterization and a mean value was calculated.
Time Frame: Three bladder scan measurements were performed immediately after each catheterization and a mean value was calculated. A maximum of 5 minutes were allowed to elapse between catheterization and bladder scan.
Population: All subjects in the investigation
Measure: Mean (Standard Deviation); unit: Residual volume in mL
Groups:
- 7 cm; 10 cm: All study participants were catheterizised with both catheters twice in a randomized order.
  Every subject is its' own control.
Arm/Group | 7 cm | 10 cm
Number analyzed (Participants) | 60 | 60
Residual volume in mL | 32.74 (41.48) | 34.78 (38.76)
Statistical Analysis 1: Comparison: 7 cm; The hypothesis that a 10 cm catheter provides equal emptying of the bladder as a 7 cm catheter was tested; Test type: Other; p = 0.8762, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Subjects With a Residual Volume >5mL or ≤5mL
Time Frame: Three bladder scan measurements were performed immediately after each catheterization and a mean value was calculated. At least 2 hours had to pass between 2 catheterizations.
Population: All subjects participating in the investigation.
Measure: Count of Participants; unit: Participants
Groups:
- 7 cm: Coloplast SpeediCath Compact catheter, 7 cm
  Four catheterizations, two with each product in a randomized order.
- 10 cm: Astra Tech POBE catheter, 10 cm
  Four catheterizations, two with each product in a randomized order.
Arm/Group | 7 cm | 10 cm
Number analyzed (Participants) | 60 | 60
Participants
  > 5 mL | 42 | 40
  ≤ 5 mL | 18 | 20
Statistical Analysis 1: Comparison: 7 cm vs 10 cm; Test type: Other; p = 0.7905, McNemar

3. Secondary Outcome: Number of Subjects With a Residual Volume >10mL or ≤10mL
Time Frame: as for outcome 1
Population: All subjecs participating in the investigation.
Measure: Count of Participants; unit: Participants
Arm/Group | 7 cm | 10 cm
Number analyzed (Participants) | 60 | 60
Participants
  >10mL | 38 | 37
  ≤10mL | 22 | 23
Statistical Analysis 1: Comparison: 7 cm vs 10 cm; Test type: Other; p = 1.00, McNemar

4. Secondary Outcome: Number of Subjects With a Residual Volume >30mL or ≤30mL
Time Frame: as for outcome 1
Population: All subjects in the investigation.
Measure: Count of Participants; unit: Participants
Arm/Group | 7 cm | 10 cm
Number analyzed (Participants) | 60 | 60
Participants
  >30mL | 19 | 26
  ≤30mL | 41 | 34

5. Secondary Outcome: Number of Subjects With a Residual Volume >50mL or ≤50mL
Time Frame: as for outcome 1
Population: All subjects participating in the investigation.
Measure: Count of Participants; unit: Participants
Arm/Group | 7 cm | 10 cm
Number analyzed (Participants) | 60 | 60
Participants
  >50mL | 15 | 16
  ≤50mL | 45 | 44

6. Secondary Outcome: Does the Subject's Bladder Feel Completely Empty After Catheterisation (All Subjects)
Description: After each catheterization the study nurse will ask the subject whether it feels as if the bladder is completely emptied or not.
  0=No and 1=Yes.
Time Frame: Question asked minutes after catheterization.
Population: All subjects participating in the investigation.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Subjects: All study participants were catheterizised with both catheters twice in a randomized order.
  Every subject is its' own control. The results of the bladder scan for cathetersization with the 7 cm long catheter minus the 10 cm long catheter shows the difference in residual volume..
Arm/Group | All Subjects
Number analyzed (Participants) | 60
score on a scale
  7 cm | 0.75 (0.40)
  10 cm | 0.83 (0.35)
  7 cm - 10 cm | -0.08 (0.26)
Statistical Analysis 1: Comparison: All Subjects; In the table 0=No and 1=Yes; Test type: Other; p = 0.0273, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: The investigation lasted for 3 months and the adverse events/adverese device effects were collected during this time.
Description: The term adverse events will be used together with the term adverse device effects in this system due to limitations in choise in reporting.
Groups:
- 7 cm: Coloplast SpeediCath Compact catheter, 7 cm Four catheterizations in total, two catheterizations with each study product in a randomized order.
- 10 cm: Astra Tech POBE catheter, 10 cm Four catheterizations in total, two catheterizations with each study product in a randomized order.
Arm/Group | 7 cm | 10 cm
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 2/60 | 1/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 7 cm (N=60) | 10 cm (N=60)
Burning sensation in urethra one hour after catheterization (Renal and urinary disorders) | 0 (0) | 1 (1) — One subject in the investigational group (10 cm catheter) reported burning sensation in urethra one hour after catheterization possibly due to the catheter. The burning sensation disappeared without any action taken.
Menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No